CLINICAL TRIAL: NCT00011050
Title: Effects of Storage on Plasma Lactate Determinations
Brief Title: Effects of Storage on Lactate in Blood Samples
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5099; AACTG A5099
Record Dates: First submitted 2001-02-09; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2004-11

CONDITIONS: HIV Infections
Keywords: Specimen Handling; Blood; Cryopreservation; Lactic Acid; Sodium Fluoride; Oxalates
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to determine whether laboratory storage of samples affects the amount of lactate over 3 years.

Lactate is a natural substance normally present in the body. Lactate levels can go up for many different reasons, including treatment with nucleotide reverse transcriptase inhibitor drugs. This study will help researchers know if stored blood samples can be used to test lactate levels.

DETAILED DESCRIPTION:
Lactic acidosis syndrome is a complication of therapy with nucleoside reverse transcriptase inhibitor (NRTI) drugs. Measurement of lactate levels is important in clinical trials of antiretroviral treatments. The preferred collection method for determining plasma lactate is with NaF/KOx tubes, while a number of ACTG studies have stored blood in ethylenediaminetetraacetic acid (EDTA) tubes. This study will analyze lactate in samples collected and stored in NaF/KOx and EDTA tubes to investigate the reliability of lactate concentrations over time.

Pre- and post-exercise blood samples are drawn from participants into NaF/KOx and EDTA tubes and a portion is tested for lactate levels immediately. The remaining portions are frozen and tested at 1, 3, 6, 12, 18, 24, and 36 months.

ELIGIBILITY:
Inclusion Criteria

Participants may be eligible for this study if they:

* Are at least 18 years old.
* Have sufficient forearm veins.

Exclusion Criteria

Participants will not be eligible for this study if they:

* Have a physical disability that prevents forearm exercise.
* Have any known medical reason, such as anemia, for not having 82 ml of blood drawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13
Dates: Start 2001-01

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dube, Study Chair; Kathleen Mulligan, Study Chair
Locations (3):
- United States (3):
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana